CLINICAL TRIAL: NCT01296477
Title: Examination of ASTHMA IQ to Improve Patient Outcomes in a Primary Care Setting
Brief Title: To Evaluate the Use of ASTHMA IQ in a Primary Care Setting
Acronym: AIQ
Status: Completed | Type: Observational
Sponsor: American Academy of Family Physicians (Other)
Collaborators: American Academy of Allergy, Asthma, and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: 10-115
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
Keywords: Asthma; ASTHMA IQ tool; Asthma Control Test (ACT); EPR-3 Guidelines, Exacerbations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Asthma IQ Primary Care Tool
- Usual Asthma Care in Primary Care

SUMMARY:
There is a mounting body of evidence suggesting that there is a large disparity between the development and the actual implementation of guideline-driven asthma care in primary and specialty care practices. To address this disparity, the American Academy of Allergy, Asthma & Immunology (AAAAI) developed a unique, comprehensive and easy-to-use Web-based tool for clinicians who treat asthma patients called "Asthma Specialist Tool to Help Manage Asthma and Improve Quality" (Asthma-IQ). This study will examine whether the use of the Asthma IQ primary care tool will improve asthma care and asthma outcomes using a randomized trial of the Asthma IQ system versus usual asthma care in the primary care setting over 1 year. At the end of 1 year, all patients will be managed using the Asthma-IQ tool for an additional year to determine if the patients managed by usual care in the first year improve when managed in conjunction with Asthma-IQ. The primary endpoint to determine if the use of the Asthma IQ tool will improve asthma patient outcomes is quarterly assessments of Asthma Control Test (ACT) scores via automated / electronic patient survey. The secondary endpoint is asthma exacerbations and there are a number of exploratory endpoints to further define the clinical utility of the primary care version of Asthma-IQ. This study will involve recruiting approximately 20 family medicine offices with approximately 20 patients each, to conduct this randomized, multiple time point intervention trial. The necessary total recruited patient sample size is 200 per group. The results of this study will help determine the utility of Web-based tools to help manage chronic diseases such as asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age 12 through 65 years at the time of screening;
2. Written informed consent obtained from the patient prior to beginning study procedures;
3. Documented clinical history of chronic persistent asthma requiring controller therapy;
4. Able to complete the study period, including follow-up period, of up to approximately 2 years; and
5. Willing to forego other forms of experimental treatment and study procedures during the study and for 30 days after the follow-up period is completed.

Exclusion Criteria:

1. History of any disease, evidence of any current disease (other than asthma), any finding upon physical examination, or any laboratory abnormality, that, in the opinion of the investigator, may compromise the safety of the patient in the study or confound the analysis of the study;
2. Lung disease other than asthma (e.g., chronic obstructive pulmonary disease, cystic fibrosis);
3. Any disease or illness, other than asthma, that is likely to require the use of systemic corticosteroids during the study period;
4. Current acute illnesses or evidence of significant active infection, such as fever ≥ 38.0°C (100.5°F) within 4 weeks of enrollment;
5. Receipt of any investigational drug therapy within 30 days or any biologic(s) within 5 half-lives prior to screening, except omalizumab for asthma;
6. Pregnancy at enrollment;
7. Breastfeeding or lactating females;
8. Elective major surgery planned from screening through study completion;
9. History of cancer other than basal cell carcinoma of the skin or cervical carcinoma-in-situ treated with apparent success with curative therapy more than 1 year prior to enrollment;
10. History of primary immunodeficiency;
11. History within the past year of excessive alcohol intake or drug addiction.
12. History of tobacco use of more than 10 pack years;
13. Plans to move from the study site area during the duration of the study.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit approximately 400 patients with chronic persistent asthma. The required sample size to identify a clinically significant difference in ACT scores from baseline and between groups requires about 200 patients per group.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
ACT scores via automated / electronic patient survey | 2 years (Surveys measured at every 3 months including baseline)

SECONDARY OUTCOMES:
Asthma exacerbations requiring the use of inhaled corticosteroids via chart reviews and automated survey | 2 years (Chart reviews performed at every 6 months and surveys measured at every 3 months including baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- AAFP National Research Network, Leawood, Kansas, United States